CLINICAL TRIAL: NCT02746900
Title: Cervical Cerclage for Preventing Spontaneous Preterm Birth in Singleton Pregnancies Without Prior Spontaneous Preterm Birth and With Short Transvaginal Ultrasound Cervical Length
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gabriele Saccone, Medical Doctor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100/16
Record Dates: First submitted 2016-04-08; First posted 2016-04-21 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth | interventions — Cerclage, Cervical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cervical cerclage (Experimental): After the woman is placed in the dorsal lithotomy position and the bladder is emptied with a urinary catheter to reduce the chance of bladder injury, surgical preparation with Betadine will be performed. Breisky retractors and Sims retractors will be used to exposure the entire cervix. Sponge ring forceps will be used to optimized visualization of the cervix and provide the necessary countertraction at the suture entry and exit sites. McDonald technique will be performed placing 4-6 bites circumferentially around the cervix. Only one stitch will be used. The suture will be places as high as feasible
  Interventions: Procedure: Cervical cerclage
- No intervention (No Intervention): Bed rest will be not recommended.

INTERVENTIONS:
Procedure: Cervical cerclage — McDonald cervical cerclage
  Arms: Cervical cerclage

SUMMARY:
Spontaneous preterm birth (SPTB) remains the number one cause of perinatal mortality in many countries, including the United States. In singleton gestations a short cervical length (CL) on transvaginal ultrasound (TVU) has been shown to be a good predictor of SPTB.

Different strategies have been adopted for prevention of SPTB. Growing interest has focused on pessary for prevention of SPTB. Cervical pessary is relatively non-invasive, easy to use, does not require anesthesia, can be used in an outpatient clinic setting, and it is easily removed when necessary. However, a recent systematic review and meta-analysis of randomized clinical trials showed that in singleton pregnancies with short cervix, prophylactic use of the pessary did not reduce the rate of spontaneous preterm delivery or improve perinatal outcome. The evidence supports the use of vaginal progesterone in singleton pregnancies with short cervix, while cervical cerclage seems to be beneficial only in the subgroup of women with both prior SPTB and TVU CL ≤25mm. Interestingly, only 235 singletons without prior SPTB,7 and 504 singletons gestations with prior SPTB,6 have been included in randomized studies on cerclage for TVU CL ≤25mm. A meta-analysis of four trials showed that cervical cerclage did not prevent SPTB in women with short TVU CL and without prior preterm birth.7 However, even if the statistical significance were not reached, they found a reduction in SPTB <35 weeks by 16% in singletons with short TVU CL and without prior SPTB (20.6% vs 31.2%; relative risk (RR) 0.84, 95% confidence interval (CI) 0.60 to 1.17) and by 24% in singletons without risk factors for SPTB (25.6% vs 33.3%; RR 0.76, 95% CI 0.52 to 1.15).

Therefore, the aim of this study is to evaluate the efficacy of cervical cerclage in prevention of SPTB in singleton pregnancies with short TVU CL in second trimester, without prior SPTB.

DETAILED DESCRIPTION:
Investigators aim to conduct a prospective, multicenter, randomized, open-label, clinical trial at Department of Reproductive Science, University of Naples Federico II. All women included in the study will provide a written informed consent to participate in the study before the randomization.

Women with TVU CL ≤25mm who will meet the inclusion criteria will be counselled by an obstetrician regarding the risk of SPTB as per standard of care. The patient will be given ample time to have all questions addressed and consider participation. If the patient agrees to participate in the study, the informed consent form will be signed and a copy will be given to the patient. Women who are eligible and consent to participate in the study will be randomly assigned to one of two groups: cervical cerclage (i.e. intervention group) or standard obstetric management (i.e. control group).

Investigators planned subgroup analyses according to different CL cutoffs (i.e. <=15 and <=10 mm); type of suture; and according to prior history of cervical surgery (i.e. LEEP or cone biopsy).

ELIGIBILITY:
Inclusion Criteria:

* 18-50 ages
* Singleton pregnancy
* Cervical length <=25mm between 18(0) and 23(6) weeks

Exclusion Criteria:

* Multiple pregnancy
* Prior spontaneous preterm birth or second trimester losses between 16(0) and 36(6) weeks
* Cerclage in situ
* Painful regular uterine contraction and/or preterm labor
* Ruptured membranes
* Major fetal defects
* Active vaginal bleeding
* Placenda previa and/or accreta
* Cervical dilation >1.5 cm and/or visible membranes by pelvic exam
* Suspicion of chorioamnionitis

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 587 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Spontaneous preterm birth (SPTB) | Less than 35 weeks gestation

SECONDARY OUTCOMES:
Spontaneous preterm birth (SPTB) | Less than 37,34,32,28 and 24 weeks gestation
Gestational age at delivery | Delivery (at birth)
  mean gestational age at delivery in weeks
Latency | Delivery (at birth)
  mean latency in days (from randomization to delivery)
chorioamnionitis | Delivery (at birth)
  chorioamnionitis histologically proven
Birth weight | Delivery (at birth)
  in grams
Admission to neonatal intensive care unit | Delivery (at birth)
respiratory distress syndrome | Delivery (at birth)
low birth weight | Delivery (at birth)
  birth weight <2500 grams
intraventricular hemorrhage | Between birth and 28 days of age
  grade 3 or 4
neonatal mortality | Between birth and 28 days of age
  death of a live-born baby within the first 28 days of life

CONTACTS AND LOCATIONS:
Locations (1):
- Gabriele Saccone, Napoli, Italy